CLINICAL TRIAL: NCT02173990
Title: A Phase 2 Study of Aflibercept and Chemotherapy as First Line Treatment for Metastatic Colorectal Cancer Assessable With DCE-US.
Brief Title: Aflibercept and Chemotherapy as First Line Treatment for Metastatic Colorectal Cancer Assessable With DCE-US (PULSAR).
Acronym: PULSAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PULSAR-1303; 2013-004540-33 (EudraCT Number)
Record Dates: First submitted 2014-02-17; First posted 2014-06-25 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: adenocarcinoma; colon and/or rectum
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aflibercept-FOLFIRI (Experimental): On day 1 of each cycle patients will receive aflibercept followed by irinotecan, 5-FU and leucovorin (FOLFIRI regimen). This treatment will be repeated every 2 weeks until RECIST progression or intolerance.
  Interventions: Drug: Aflibercept-FOLFIRI

INTERVENTIONS:
Drug: Aflibercept-FOLFIRI — Aflibercept : 4 mg/kg, IV over 1 h on Day 1
  FOLFIRI :
  * Irinotecan 180 mg/m² IV infusion in 500 mL D5W (5% Dextrose in Water solution) over 90 minutes and dl leucovorin* 400 mg/m² IV infusion over 2 hours, at the same time, in bags using a Y-line, followed by :
  * 5-FU 400 mg/m² IV bolus given over 2-4 minutes, followed by :
  * 5-FU 2400 mg/m² continuous IV infusion in 500 mL over 46-hours.
    * *400 mg/m² of leucovorin expressed in dl racemic. When the l-isomer form is used the dose should be divided by 2, i.e. 200 mg/m²
  Other Names: ZALTRAP-FOLFIRI

SUMMARY:
The PULSAR trial is an international, investigator-initiated, single arm open-label phase II study. The aim of this study is to measure the clinical activity of the combination FOLFIRI-aflibercept in an homogeneous group of patients with metastatic colorectal cancer, and treated with a FOLFIRI-aflibercept regimen as first line treatment.

DETAILED DESCRIPTION:
Patients with an unresectable metastatic colorectal carcinoma (mCRC) histologically proven will be treated with a combination of Irinotecan/bolus-infusion-5-Fluorouracil/Leucovorin (FOLFIRI regimen) and aflibercept. On day 1 of each cycle patients will receive aflibercept followed by irinotecan, 5-Fluorouracil (FU) and leucovorin (FOLFIRI regimen). This treatment will be repeated every 2 weeks until RECIST progression or unacceptable toxicities, investigator's decision or patient's refusal of further treatment or death, whichever comes first.

All patients will be assessed during their FOLFIRI-aflibercept with Dynamic Contrast Enhanced Ultrasound (DCE-US) at baseline, D7 (± 1 day), D28 (± 2 days).

The recruitment period is 24 months. The average duration of the study per patient will be approximately 12 months, i.e. 3 weeks for screening, 10 months for the combination of FOLFIRI plus aflibercept and 30 days for follow-up of adverse events after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent, and willing and able to comply with protocol requirements
2. Histologically proven adenocarcinoma of the colon and/or rectum
3. Metastatic disease confirmed clinically/radiologically, and evaluable by dynamic contrast ultrasound
4. No prior therapy for metastatic disease
5. Duly documented inoperable metastatic disease, i.e. not suitable for complete curative surgical resection
6. At least one measurable or evaluable lesion as assessed by CT-scan or MRI (Magnetic Resonance Imaging) according to RECIST v1.1
7. Age ≥ 18 years
8. Eastern Cooperative Oncology Group (ECOG) Performance status (PS) 0-2
9. Adequate hematological status: neutrophils (ANC) ≥ 1.5 x109/L; platelets ≥ 100x109/L; haemoglobin ≥ 9g/ dL
10. Adequate renal function: serum creatinine level < 1.5 mg/dl and Glomerular Filtration Rate > 50 ml/min by cockroft/ Gault formula
11. Adequate liver function: serum bilirubin ≤ 1.5 x upper normal limit (ULN), alkaline phosphatase, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) < 5 x ULN
12. Proteinuria < 2+ (dipstick urinalysis) or ≤ 1g/24 hour
13. Female patients must commit to using reliable and appropriate methods of contraception until at least 6 months after the end of Aflibercept and 3 months after the end of Irinotecan (when applicable). Male patients with a partner of childbearing potential must agree to use contraception in addition to having their partner use another contraceptive method until at least 6 months after the end of Aflibercept and 3 months after the end of Irinotecan.

Exclusion Criteria:

1. Uncontrolled hypercalcemia
2. Uncontrolled systemic hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg despite medical therapy), or history of hypertensive crisis, or hypertensive encephalopathy
3. Right-left shunt or severe pulmonary arterial hypertension (pulmonary artery pressure > 90 mmHg)
4. Respiratory distress syndrome
5. Concomitant antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy)
6. Treatment with any other investigational medicinal product within 28 days prior to study entry
7. History or presence of Central Nervous System (CNS) metastasis unless adequately treated (e.g. non irradiated CNS metastasis, seizures not controlled with standard medical therapy)
8. Gilbert's syndrome
9. Intolerance to atropine sulfate or loperamide
10. Known dihydropyrimidine dehydrogenase deficiency
11. Treatment with Cytochrome P450 3A4 (CYP3A4) inducers unless discontinued > 7 days prior to registration
12. Any of the following in 3 months prior to inclusion: grade 3-4 gastrointestinal bleeding (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or chronic inflammatory bowel disease, or diverticulitis
13. Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for > 5 years,
14. Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 days
15. Pregnant or breastfeeding women
16. Patients with known allergy to any excipients to study drugs (including hypersensitivity to sulphur hexafluoride or to any of the components of SonoVue)
17. History of myocardial infarction and/or stroke or other arterial thrombotic events or pulmonary embolism or unstable angina pectoris within 6 months prior to registration
18. Poorly controlled cardiac arrhythmias
19. Typical Angina Pectoris at rest within the previous 7 days, or significant worsening of cardiac symptoms in the previous 7 days, or recent intervention on the coronary arteries or other factors suggesting clinical instability (eg recent deterioration of ECG changes in clinical parameters or biological), or acute heart failure, or heart failure stage III or IV, or severe arrhythmias
20. Bowel obstruction
21. History of severe tumour bleeding or bleeding disorders
22. Poorly controlled anti-coagulation therapy (INR > 3.0 on coumadin or heparin compounds)
23. Palliative radiation therapy within 4 weeks prior to registration
24. St John's Wort medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Progression-Free Rate will be assessed according to RECIST 1.1 with central radiological review. | At 10-month

SECONDARY OUTCOMES:
Overall Response Rate (ORR) will be determined according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. | through the end of study treatment, an average of 1 year
Best Response Rate (BRR) | through the end of study treatment, an average of 1 year
Progression-free survival (PFS) | through study completion, an average of 3 years
Progression-free survival rate | through study completion, an average of 3 years
Patterns of PFS according to DCE-US early assessment | at day 28 ± 2
Pharmacodynamic activity | at day 7 ± 1, and day 28 ± 2
Safety and tolerance | up to 30 days after the end of the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ADENIS, MD, PhD, Study Director — Centre Oscar Lambret - France
Locations (8):
- France (8):
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Kremlin Bicetre, Le Kremlin-Bicêtre
  - Centre Oscar Lambret, Lille
  - CHRU, Lille
  - Institut Paoli Calmettes, Marseille
  - Hôpital Universitaire Paul Brousse, Villejuif
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No